CLINICAL TRIAL: NCT00804414
Title: A Randomised, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Soluble Beta-1,3/1,6-glucan (SBG) in Chronic Foot Ulcers in Patients With Diabetes
Brief Title: Efficacy and Safety Study of Soluble Beta-1,3/1,6-glucan (SBG) Versus Placebo in Chronic Diabetic Foot Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotec Pharmacon ASA (Industry)
Responsible Party: Vice President Clinical Development, Biotec Pharmacon ASA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBG-1-13
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes; Diabetic Ulcer
Keywords: Diabetes; Diabetic ulcer; Chronic ulcer; SBG
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: SBG
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: SBG — Solution for topical use
  Arms: 1
Drug: Placebo Comparator — Solutin for topical use
  Arms: 2

SUMMARY:
Evaluation of efficacy and safety of SBG vs placebo in the treatment of chronic diabetic foot ulcers.

DETAILED DESCRIPTION:
The objective of this study is to evaluate efficacy and safety of soluble beta-1,3/1,6-glucan (SBG) on chronic diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic diabetic foot ulcer

Exclusion Criteria:

* Insufficient nutritional status, renal function or diabetes control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Compare the proportion of patients in the two arms who have complete healing of target ulcer | Maximum 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain